CLINICAL TRIAL: NCT02389972
Title: Effectiveness of Dasatinib(Sprycel®) in Adult Patients With Chronic Myeloid Leukemia in China: A Multicenter, Registry Study
Brief Title: Effectiveness of Dasatinib in Adult Patients With Chronic Myeloid Leukemia in China: A Multicenter, Registry Study
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA180-518
Record Dates: First submitted 2014-10-29; First posted 2015-03-17 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Leukemia, Myelogenous, Chronic, BCR-ABL Positive
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CML patients treated with dasatinib: Cohort of chronic myeloid leukemia patients treated with second-line dasatinib (Sprycel)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib
  Other Names: Sprycel

SUMMARY:
The primary objective is to describe the effectiveness of dasatinib (Sprycel®) in CML patients in China in the real-world clinical practice setting.

DETAILED DESCRIPTION:
Breakpoint cluster region (BCR)

Abelson murine leukemia viral oncogene homolog 1 (c-ABL)

Chronic myeloid leukemia (CML)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

Because this is a product registry study, it will include adult CML patients in any phase treated with dasatinib in China if they meet the following criteria:

* Willing and able to provide written informed consent
* ≥18 years of age
* Confirmed diagnosis of CML patients by attending physician
* Naive to dasatinib before enrollment in study treatment or have received <3 months of dasatinib treatment
* Plan to or are receiving dasatinib therapy based on physician's clinical judgment
* Administered dasatinib after imatinib-resistance or intolerance

Exclusion Criteria:

- Patients participating in clinical trials for CML that explicitly prohibit recruitment in additional studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be naive to dasatinib before the enrollment period, be over the age of 18 years with a confirmed diagnosis of any phase CML by the treating physician, and are to initiate treatment with dasatinib based on the physician's clinical judgement
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2013-04-11 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Rate of Hematologic response (HR) for Chronic phase (CP), Advanced phase (AP),Blast phase (BP) | Upto 2 years
  Hematological Response is a normalization of the blood counts, particularly white blood cell counts. This is the first noticeable indicator that treatment is beginning to work, though not necessarily in the bone marrow
Rate of Cytogenetic response (CR) for Chronic phase, Advanced phase,Blast phase | Upto 2 years
  Cytogenetic Response is a response to treatment of CML that occurs in the marrow, rather than just in the blood
Rate of Molecular response (MR) for Chronic phase,Advanced phase,Blast phase | Upto 2 years
  Molecular response is defined as no detectable BCR-ABL observed through Quantitative polymerase chain reaction (Q-PCR) (International Scale) using an assay with a sensitivity of at least 4.5 logs below the standardized baseline

SECONDARY OUTCOMES:
Demographic and baseline characteristics of patients using dasatinib including health insurance, concomitant regimens, risk scores, and comorbidities based on patient-reported questionnaire | Upto 2 years
  Type and percentage of each variable: health insurance, concomitant regimens and comorbidities; patients distribution by Sokal score
Dasatinib treatment pattern, including medication adherence and treatment interruption based on patient-reported questionnaire | Upto 2 years
  Dasatinib starting dose and administration schedule, cumulative dose, maximum daily dose and duration of exposure; dose alterations (including changes in frequency, reductions and or delays) and reason(s) for dose alterations; discontinuation and reason(s) for dasatinib discontinuation
Relationship between time to initiation of dasatinib after imatinib failure and best response to dasatinib | Upto 2 years
Progression-free survival (PFS) | Upto 2 years
Overall survival (OS) | Upto 2 years
Safety of dasatinib measured by incidence and severity of adverse events | Upto 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Wuhan, Hubei, China

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx